CLINICAL TRIAL: NCT05954416
Title: National Cohort for Evaluation of the Burden of Rare Skin Diseases
Brief Title: FARD (RaDiCo Cohort) (RaDiCo-FARD)
Acronym: FARD
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-78
Record Dates: First submitted 2023-06-26; First posted 2023-07-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Inherited Epidermolysis Bullosa; Ichthyosis; Ectodermal Dysplasia; Incontinentia Pigmenti; Neurofibromatosis Type 1; Albinism; Pemphigus; Mucous Membrane Pemphigoid; Palmoplantar Keratoderma
MeSH Terms: conditions — Ichthyosis; Ectodermal Dysplasia; Incontinentia Pigmenti; Neurofibromatosis 1; Albinism; Pemphigus; Pemphigoid, Benign Mucous Membrane; Keratoderma, Palmoplantar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to conduct a prospective assessment of the individual Burden of 9 rare skin diseases to assess disability in the broadest sense of the term (psychological, social, economic and physical) for patients and/or families.

Two types of indicators will be used to reach this objective :

1. an individual burden score calculated based on a burden questionnaire created specifically, approved and designed to understand the tendency to changes in care and lifestyles. The burden questionnaire should be used by patients and/or their family themselves in self-assessment.
2. a descriptive analysis of all resources (medical and non-medical) used by the family unit to manage the disease.

ELIGIBILITY:
Inclusion criteria :

* adults or children with a confirmed diagnosis of one of the 9 following rare skin disease: Inherited epidermolysis bullosa, Ichthyosis, Ectodermal dysplasia, Incontinetia Pigmenti, Neurofibromatosis type 1, Albinism, Pemphigus, Mucous membrane pemphigoid or Palmoplantar keratoderma.
* prevalent or incident and followed in one the reference/competence centers of the FIMARAD healthcare network,
* able to understand a survey (for child, survey should be understood by parents),
* having given their signed consent to participate to the cohort RaDiCo-FARD (parents' consent for child).

Non-inclusion criteria :

* Patients, for whom regular care follow-up is not feasible with the FIMARAD healthcare network sites,
* Unconfirmed diagnosis (according to criteria for each disease),
* Patients (and/or parents) not able to understand a survey
* Patients (and/or parents) not having given their signed consent to participate to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study concerns patients affected by one the 9 following rare skin diseases: Inherited epidermolysis bullosa, ichthyosis, ectodermal dysplasia, Incontinentia Pigmenti, neurofibromatosis type 1, albinism, pemphigus, mucous membrane pemphigoid, and palmoplantar keratoderma recruited and followed in a reference/competence centre of the healthcare network of rare dermatologic diseases, FIMARAD.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2027-03-07 (Estimated); Study Completion 2027-03-07 (Estimated)

PRIMARY OUTCOMES:
Individual burden score for each selected rare disease | Through study completion, an average of 5 years
  Before 16 years old, we will focus on the burden of families. After 16 years old, the patient's parent will continue to answer to the family Burden questionnaire and the patient will start to answer to the adult's Burden questionnaire.

SECONDARY OUTCOMES:
Description of calculated scores based on widely used survey completed by patients | Through study completion, an average of 5 years
Description of calculated scores based on widely used survey completed by parents | Through study completion, an average of 5 years
Description of variations of quality-of-life scores. | Through study completion, an average of 5 years
Validation of the clinical severity score for disease which have none at the beginning of the study and description of clinical severity score. | Through study completion, an average of 5 years
Descriptive analysis of the socio-economic Burden. | Through study completion, an average of 5 years
Descriptive analysis of the Individual Health Care Cost. | Through study completion, an average of 5 years
Search for association between individual burden score and clinical severity of the disease. | Through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine BODEMER, Principal Investigator — INSERM UMR 1163
Locations (14):
- France (14):
  - Hôpital Avicenne, Bobigny
  - Hôpital des Enfants - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital Henri-Mondor, Créteil
  - Hôpital François Mitterrand, Dijon
  - Hôpital Dupuytren, Limoges
  - Hôpital de la Timone, Marseille
  - Hôpital Saint-Eloi, Montpellier
  - Hôpital l'Archet, Nice
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Robert-Debré, Reims
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Larrey, Toulouse
  - Hôpital Trousseau, Tours